CLINICAL TRIAL: NCT03242460
Title: The Safety and Efficacy of Pomalidomide in Combination With Cyclophosphamide and Dexamethasone (PCD) in the Transplant-ineligible Patients With Relapsed and/or Refractory Multiple Myeloma (MM) Who Had Lenalidomide Plus Dexamethasone (LD) Following Frontline Bortezomib Combined Chemotherapy, Open-labeled, Multicenter Phase II Study
Brief Title: The Safety and Efficacy of Pomalidomide in Combination With Cyclophosphamide and Dexamethasone (PCD) in the Transplant-ineligible Patients With Relapsed and/or Refractory Multiple Myeloma (MM)
Acronym: PORYOU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kosin University Gospel Hospital (Other)
Responsible Party: Principal Investigator, Ho Sup Lee, MD, PhD. associate professor, Division of hematology-Oncology, Kosin University Gospel Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PORYOU
Record Dates: First submitted 2017-08-01; First posted 2017-08-08 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Relapsed and/or refractorY Multiple Myeloma
MeSH Terms: interventions — pomalidomide; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: the transplant-ineligible patients with Relapsed and/or refractorY multiple myeloma (MM) who had lenalidomide+dexamethasone (LD) following frontline bortezomib combined chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pomalidomide, Dexamethasone, Cyclophosphamide (Experimental): Pomalidomide 4mg Days 1-21 Dexamethasone 20mg Days 1, 8, 15, 22 Cyclophosphamide 400mg Days 1, 8, 15
  Interventions: Drug: Pomalidomide 4 MG; Drug: Dexamethasone 20mg; Drug: Cyclophosphamide 400mg

INTERVENTIONS:
Drug: Pomalidomide 4 MG — Pomalidomide 4mg Days 1-21
  Other Names: pomalyst
Drug: Dexamethasone 20mg — Dexamethasone 20mg Days 1, 8, 15, 22
Drug: Cyclophosphamide 400mg — Cyclophosphamide 400mg Days 1, 8, 15

SUMMARY:
In Korea, VMP is most commonly used as frontline treatment in patients with newly diagnosed MM who were ineligible for high-dose therapy. Recently National Insurance began to reimburse the second-line LD when the bortezomib-containing treatment failed to salvage the patients. Patients who have relapsed MM after exposure to the above agents and have progressive disease have a short life expectancy. Third-line therapy is needed for retrieving the patients hereafter. And substantial proportion of patients will attain an advanced age. To examine if time to disease progression is maintained and tolerability is improved with lower dexamethasone dose, the dose of dexamethasone is reduced when at least a minimal response is achieved after 3 months of treatment with the initial dose. Three months later (6 months after the initial treatment), the response remains in stable disease, 2nd dose reduction (dexamethasone 10mg or prednisone 50mg) will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have evaluable multiple myeloma with at least one of the following (within 21 days of starting treatment)

  * Serum M-protein ≥ 0.5g/dL, or
  * In subjects without detectable serum M-protein, Urine M-protein ≥ 200mg/24 hour, or serum free light chai (sFLC) > 100mg/L (involved light chain) and an abnormal kappa/Lambda ratio
* Patients were ineligible for autologous stem cell transplantation
* Must be relapse refractory to initial therapy with bortezomib, melphalan and prednison and then lenalidomide plus dexamethasone.
* Refractoriness is defined as disease progression on treatment or progression within 6 months after the last dose of a given therapy. Relapse is defined according to the criteria of IMWG
* Males and females ≥ 18 years of age or > country's legal age for adult consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
* Patients must meet the following clinical laboratory criteria with 21 days of starting treatment:

  * Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet ≥ 50,000/mm3 (≥ 30,000/mm3 if myeloma involvement in the bone marrow is >50%)
  * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
  * Calculated creatinine clearance ≥ 30mL/min or creatinine < 3mg/dL.
* Written informed consent in accordance with federal, local and institutional guidelines

Exclusion Criteria:

* Female patients who are lactating or pregnant
* Multiple Myeloma of IgM subtype
* Glucocorticoid therapy (prednisolone > 30mg/day or equivalent) within 14 days prior to informed consent obtained
* POEMS syndrome, plasma cell leukemia or circulating plasma cells ≥ 2 x 109/L, Waldenstrom's Macroglobulinaemia, or Patients with known amyloidosis
* Peripheral neuropathy grade > 2
* Chemotherapy with approved or investigation anticancer therapeutics within 21 days prior to starting pomalidomide treatment
* Focal radiation therapy within 7 days prior to start of pomalidomide. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to start of pomalidomide
* Immunotherapy (excluding steroids) 21 days prior to start of pomalidomide
* Major surgery (excluding kyphoplasty) within 28 days prior to start of pomalidomide
* Active congestive heart failure (New York Heart Association [NYHA] Class III or IV), symptomatic ischaemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 4 months prior to informed consent obtained
* Known HIV seropositive, hepatitis C infection, and/or hepatitis B (except for patients with hepatitis B surface antigen or core antibody receiving and responding to antiviral therapy directed at hepatitis B: these patients are allowed)
* Second malignancy within the past 3 years except:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Breast carcinoma in situ with full surgical resection
* Patients with steroid or lenalidomide hypersensitivity
* Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to starting pomalidomide treatment
* Any clinically significant medical disease or psychiatric condition that, in the investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-05-12; Primary Completion 2019-04-24 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Median Progression-free Survival (PFS) | 2 years follow up
  Kaplan-Meier method

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years follow up
  International Myeloma Working Group,( IMWG)
Overall survival (OS) | 2 years follow up
  Kaplan-Meier method
Safety evaluations assessed using Common Terminology Criteria for Adverse Events v4.0 | 2 years follow up
  Common Terminology Criteria for Adverse Events v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic university of korea, Seoul ST. Mary's Hospital., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
KMMWP